CLINICAL TRIAL: NCT05410899
Title: Investigation of Effectiveness of Pelvic Floor Health Education and Exercise Program Effectiveness on Women With Urinary Incontinence
Brief Title: Exercise and Pelvic Floor Health Education Program Effectiveness
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, SEVGİ GAMZE İRİ, Msc Physiotherapist, Harran University
Other Study IDs: Harran üniversitesi
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Urinary Incontinence; Pelvic Floor Disorders; Exercise Addiction
Keywords: urinary incontinence; exercise; pelvic floor; health education
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders; Motor Activity; Health Education | interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pelvic Floor Health Education: Education will compose presentation about women health, urinary incontinence, teaching anatomy of the pelvic floor and bladder training
  Interventions: Other: exercise
- Pelvic Floor Health Education and Exercise Program: pelvic floor health education and exercise of pelvic floor muscles for 12 weeks
  Interventions: Other: exercise
- Control: This goup will continue routine treatment such as medication usage
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Women with urinary incontinence will done exercise including pelvic floor muscle and will taught pelvic floor muscle anatomy, physiology, disorders, treatment of disease
  Other Names: pelvic floor health education

SUMMARY:
The aim of the study is investigation of the effectiveness of Pelvic Floor Health Education and exercise program in women with Urinary Incontinence. Women diagnosed with both stress and mixed type urinary incontinence were included the study. Pelvic Floor Health Education and exercise program were applied to women for 12 weeks.

DETAILED DESCRIPTION:
3 group were created; the first group will applied Pelvic floor health education composed presentation about women health,urinary incontinence, teaching anatomy of the pelvic floor and bladder training ,second group will applied both pelvic floor health education and exercise of pelvic floor muscles for 12 weeks and third group will be control group.Women with urinary incontinence were included the study are continued 12 weeks . First evaluation is done before education and exercise program, and second evaluation in 6.week and last evaluation after 12 weeks exercise and education program.

ELIGIBILITY:
Inclusion Criteria:

1. The ages between 18-65 with urinary incontinence
2. Volunteer women who can regularly apply the Pelvic floor muscle exercise program

Exclusion Criteria:

1. Having pelvic organ prolapse (Stage≥2),
2. Women who are in the neonatal and postnatal period (up to 3 months after birth),
3. Situations that will prevent evaluation or communication (cognitive problems, etc.).
4. Having a neurological disorder,having urinary tract infection,
5. Those who received urinary incontinence treatment or had an operation, • Women who have received training on the pelvic floor before

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Urinary incontinence is more common in women than men
Study Population: The ages between 18 -65 women with urinary incontinence, applying pelvic floor muscle exercise
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2022-06-04 (Actual); Primary Completion 2022-09-26 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Incontinence severity | 3 month
  urinary incontinence severity changes frequency of incontinence, using Sandvik severity scale quantity of incontinence, type and time of incontinence, also using voiding diary for three days composed of fluid intake time, voiding time, urinary incontinence time and amount

SECONDARY OUTCOMES:
Life style | 3 month
  women with urinary incontinence decrease quality of life,using visual analog scale (VAS) isolation from their environment, trouble with family

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University Hospital, Sanliurfa, Turkey/Şanlıurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No